CLINICAL TRIAL: NCT06551051
Title: A Single-arm Phase II Study of Duloxetine for the Treatment of Neurotoxicity Induced by Antibody-drug Conjugate
Brief Title: ADC-induced Neurotoxicity Treated With Duloxetine
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Hongxia Wang, professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIPN-ADC-001
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Solid Tumour
Keywords: ADC; Neurotoxicity; Duloxetine
MeSH Terms: conditions — Neurotoxicity Syndromes | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- duloxetine (Experimental): Patients were treated with duloxetine at a recommended dose of 40mg/day, increasing to a maximum dose of 60mg/day after seven days of non-significant discomfort.
  Interventions: Drug: duloxetine

INTERVENTIONS:
Drug: duloxetine — Patients were treated with duloxetine at a recommended dose of 40mg/day, increasing to a maximum dose of 60mg/day after seven days of non-significant discomfort.
  Other Names: duloxetine hydrochloride

SUMMARY:
RATIONALE: Duloxetine may lessen peripheral neuropathy caused by chemotherapy. It is not yet known whether duloxetine is effective in treating peripheral neuropathy caused by antibody-drug conjugate.

PURPOSE: This single arm phase II trial is studying duloxetine to see how well it works in treating peripheral neuropathy caused by antibody-drug conjugate in patients with cancer.

DETAILED DESCRIPTION:
This study is a single arm phase II study. The study consisted of a screening period (subjects signed informed consent up to no more than 28 days before the first treatment of the study), a treatment period (treatment termination was defined as termination of treatment for any reason, such as imaging confirmation of disease progression, intolerance of toxicities despite dose adjustments, or early withdrawal for any reason), and a follow up period (consisting of an end-of-treatment visit, a safety visit, and a survival follow up).

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥ 18 years;
2. patients with a diagnosis confirmed by histological and/or cytological examination combined with imaging or ultrasound assessment of various advanced cancers;
3. consent to treatment;
4. ECOG score: 0 to 2;
5. have a recent treatment regimen that includes an ADC class of drug and experience a resulting grade 2 or higher peripheral neurotoxicity that has been discontinued, and grade 2 or higher peripheral neurotoxicity that has lasted for more than 28 days; and the tumour remains stable in the short term, and may be treated without the use of drugs that can cause peripheral neurotoxicity (ADCs, platinums, paclitaxels, etc.) for a period of two months.
6. Have adequate organ function:

(1) blood routine: Absolute Neutrophil Count (ANC) 1.5×109/L, Platelet (PLT) ≥70×109/L, Hemoglobin (HGB) ≥80g/L; (2) Liver function: serum Total Bilirubin (TBIL) ≤1.5×Upper Limit of Normal Value (ULN); Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≥1.5×Upper Limit of Normal Value (ULN). Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≤3×ULN; serum albumin ≥28 g/L; Alkaline Phosphatase (ALP) ≤5×ULN; after routine hepatoprotective treatment meeting the above criteria, and can be stabilised for at least 1 week after evaluation by the investigator can be enrolled; 3) Renal function: serum creatinine (Cr) ≤ 2 × ULN or creatinine clearance ≥ 30 mL/mi (applying the standard Cockcroft-Gault formula); 7. a predicted survival of ≥ 3 months; and tumour stability in the near future. 8. ability to comply with study visit schedules and other protocol requirements.

Exclusion Criteria:

1. peripheral neurotoxicity of grade 2 or higher has occurred with platinum-containing paclitaxel chemotherapy prior to prior ADC class administration, and the toxicity has not significantly worsened before or after ADC administration;
2. patients with severe diabetes mellitus and peripheral vascular disease;
3. patients with a history of neuropathy due to any type of nerve compression (e.g., carpal tunnel or tarsal tunnel syndrome, radiculopathy, spinal stenosis, brachial plexopathy), severe depression, suicidal ideation, bipolar disorder, alcoholism, and severe eating disorders
4. active or uncontrolled serious infections (≥ CTCAE grade 2 infections) requiring administration of systemic antibacterial, antifungal or antiviral therapy, including tuberculosis infections.
5. active hepatitis (aminotransferases do not meet the inclusion criteria, Hepatitis B reference: HBV DNA ≥2000 IU/ml or ≥104 copy number/ml; Hepatitis C reference: HCV RNA ≥2000 IU/ml or ≥104 copy number/ml; below the above criteria after nucleoside analogue antiviral therapy, can be enrolled); Chronic Hepatitis B viral carriers with HBV DNA < 104 IU/ml, must receive concomitant antiviral therapy during the trial to be enrolled;
6. renal failure requiring haemodialysis or peritoneal dialysis;
7. those with a history of immunodeficiency, including being HIV-positive or suffering from other acquired or congenital immunodeficiency diseases, or with a history of organ transplantation
8. those with severe nausea, headache, insomnia, fatigue, drowsiness, dry mouth, dizziness and constipation
9. those with a history of active tuberculosis
10. uncontrolled, still need repeated drainage appearing ascites, pericardial effusion, pleural effusion;
11. research treatment related:
12. patients who have undergone major organ transplantation
13. those who have undergone major surgical treatment, incisional biopsy, or significant traumatic injury within 28 days prior to the start of study treatment; or those who have longstanding unhealed wounds or fractures
14. those who have experienced a severe hypersensitivity reaction following the use of monoclonal antibodies; those with known hypersensitivity to active ingredients or excipients such as the study drug;
15. those who are participating or have participated in other clinical studies within 4 weeks prior to the start of the study
16. those with a history of severe allergy
17. have a risk of bleeding, or coagulation disorders, or are receiving thrombolytic therapy
18. have a history of psychotropic substance abuse that is not amenable to cessation or have a psychiatric disorder
19. subjects with concomitant medical conditions that, in the judgement of the investigator, seriously jeopardise the safety of the subject or interfere with the completion of the study, or who are considered otherwise unsuitable for enrolment subjects who, in the judgement of the investigator, have concomitant medical conditions that, in the judgement of the investigator, seriously jeopardise the safety of the subject or interfere with the completion of the study, or who are considered otherwise unsuitable for enrolment. Past history of definite neurological and psychiatric disorders such as dementia, epilepsy, or seizure proneness
20. in the judgement of the Investigator, a concomitant medical condition (e.g., severe diabetes mellitus, thyroid disease, psychiatric illness, etc.) which is a serious risk to the safety of the subject or which interferes with the subject's ability to complete the study, or the presence of a serious and/or unstable medical, psychiatric, or other condition (including abnormalities in laboratory tests) which interferes with the safety of the patient or with the patient's ability to provide informed consent, or any psychological, family, sociological, or psychological condition which interferes with the study protocol and the follow-up plan. Psychological, familial, sociological, or geographic conditions that affect the study protocol and follow-up plan that the investigator deems unsuitable for participation in this clinical trial for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity subscale | Day0 and Day36
  FACT-GOG-NTx scale neurotoxicity score (duloxetine treatment day 0 and 36) (4-point decrease in neurotoxicity score).
  The FACT-GOG-NTx scale, is a tool used to assess the symptoms of chemotherapy-induced peripheral neuropathy (CIPN). This scale consists of 11 items, each item is scored on a 5-point scale (0=not at all, 4=very much), with a higher total score indicating more severe CIPN symptoms.
  In the study, the Minimal Clinically Important Difference (MCID) for the FACT-GOG-NTx scale was estimated to be between 1.38 and 3.68, which means that changes within this range are considered to be clinically meaningful.
  FACT/GOG-NTx provides a targeted assessment of symptoms of peripheral neuropathy, including sensory, motor, and auditory problems and cold sensitivity.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 16 months
  Adverse events (AEs), including type, incidence, grading (based on NCI-CTCAE V5.0 criteria), severity, duration, and relevance to the study medications.
Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity subscale | 3 months
  The FACT-GOG-NTx scale, is a tool used to assess the symptoms of chemotherapy-induced peripheral neuropathy (CIPN). This scale consists of 11 items, each item is scored on a 5-point scale (0=not at all, 4=very much), with a higher total score indicating more severe CIPN symptoms.
  In the study, the Minimal Clinically Important Difference (MCID) for the FACT-GOG-NTx scale was estimated to be between 1.38 and 3.68, which means that changes within this range are considered to be clinically meaningful.
  FACT/GOG-NTx provides a targeted assessment of symptoms of peripheral neuropathy, including sensory, motor, and auditory problems and cold sensitivity.
Numerical rating scale | Day0 and Day36
  A numeric pain rating scale is a single-item question that asks the patient to rate his or her pain on a scale of 0 to 10, using the anchors of "no pain" and "worse pain imaginable."
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | Day0 and Day36
  Minimum Value: 0 (indicating the best possible health state) Maximum Value: 100 (indicating the worst possible health state) Higher scores indicate a worse quality of life or more severe symptoms. The scale includes both multi-item scales and single items to reflect various aspects of health-related quality of life.
  The scale consists of 30 questions measuring the patient's quality of life in terms of five functions (physical, daily living, cognitive, emotional and social), three symptoms (fatigue, pain, nausea and vomiting), and overall health, overall quality of life, and six other separate items (quality of sleep, appetite, diarrhoea, constipation, respiratory distress, and economic status).
Neurotoxicity score assessed by CTCAE 5.0 scale | Day0 and Day36
  Grade 1: asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated
  Grade 2: moderate; minimal, local or noninvasive intervention indicated; limiting age appropriate instrumental activities of daily living
  Grade 3: severe or medically significant but not immediately life threatening; hospitalisation or prolongation of existing hospitalisation indicated; disabling; limiting self care activities of daily living
  Grade 4: life threatening consequences; urgent intervention indicated

CONTACTS AND LOCATIONS:
Overall Officials: Hongxia Wang, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No